CLINICAL TRIAL: NCT01966523
Title: A Pilot Study of an RCT to Improve Infection Management in Advanced Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susan Mitchell, MD, Senior Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NIH R21AG042325
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2015-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Provider Training: i. on-line education course and ii. algorithms and checklists. The course consists of 4 cases: 2 for urinary tract infection and 2 for lower respiratory tract infections with multiple choice questions and evidence-based feedback. To reinforce provider learning, posters displaying algorithms guiding appropriate antimicrobial initiation for infections will be placed in all nursing home units. Laminated pocket cards with the algorithms will be given to providers. Providers will complete simple checklists for each suspected infection throughout the study. B. Proxy Information: The printed material explains, in a lay fashion: i. the nature of infection in advanced dementia, ii. treatment options, iii. concerns about antimicrobial overuse, and iv. features of appropriate antimicrobial use.
  Interventions: Behavioral: Intervention
- Usual Care (Other): Residents will receive usual care for infections
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention — Provider Training: i. on-line education course and ii. algorithms and checklists. The course consists of 4 cases: 2 for urinary tract infection and 2 for lower respiratory tract infections with multiple choice questions and evidence-based feedback. To reinforce provider learning, posters displaying algorithms guiding appropriate antimicrobial initiation for infections will be placed in all nursing home units. Laminated pocket cards with the algorithms will be given to providers. Providers will complete simple checklists for each suspected infection throughout the study. B. Proxy Information: The printed material explains, in a lay fashion: i. the nature of infection in advanced dementia, ii. treatment options, iii. concerns about antimicrobial overuse, and iv. features of appropriate antimicrobial use.
  Other Names: Infection Management Practice Intervention
  Arms: Intervention
Other: Control
  Arms: Usual Care

SUMMARY:
To conduct a pilot study of cluster randomized clinical trial of an practice intervention to improve the quality of care for suspected lower respiratory and and urinary tract infections among 60 nursing home residents with advanced dementia living in 4 facilities (2 matched intervention/control pairs) for 12 months. We hypothesize that 1. In the intervention compared to the control facilities there will be a trend towards a greater proportion of infections for which antimicrobials were initiated appropriately, and 2. in the intervention compared to the control facilities there will be a trend towards higher proxy satisfaction with decision-making, fewer hospital transfers, and lower antimicrobial exposure.

ELIGIBILITY:
Inclusion Criteria:

Resident eligibility criteria include: 1) Age > 65, 2) Dementia, 3) Global Deterioration Scale score of 7,59 and 4) a proxy is available who can speak in English. Features of Global deterioration stage 7 include: profound memory deficits (cannot recognize family), total functional dependence, speech < 5 words, incontinence, and inability to ambulate.

Eligibility criteria for providers in the intervention nursing homes include: Medical Doctor,a. nurse, nurse practitioner, physician assistant identified by a senior administrator as an individual who cares for residents with advanced dementia, and is 2. able to communicate in English because on-line course and algorithms are in English., and 3. over 21 years of age.

-

Exclusion Criteria:

Residents with cognitive impairment due to causes other than dementia (e.g., head trauma) and in short-term, sub-acute SNFs will be excluded. -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
proportion of suspected infectious episodes for which antimicrobials were initiated appropriately | 12 months
  The primary outcome will be the proportion of suspected infectious episodes for which antimicrobials were initiated appropriately defined by 2 factors: i. minimal clinical criteria to start antimicrobials are met based on consensus guidelines, ii. treatment was consistent with proxy preferences (based on proxy interview).

SECONDARY OUTCOMES:
hospital transfers | 12 months
  proportion of episodes for which residents were transferred to the hospital,

OTHER OUTCOMES:
antimicrobial use | 12 months
  total antimicrobial use among residents defined as days of therapy per 1000 resident-days
Decision satisfaction | 12 months
  proxy satisfaction with decision-making as measured by the Decision Satisfaction Index,

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew SeniorLife, Boston, Massachusetts, United States